CLINICAL TRIAL: NCT03052790
Title: Comparison of Implant Positioning With Robotic Aided Surgery and Traditional Jig Positioning in Total Knee Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Adam M Freedhand, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-16-1096
Record Dates: First submitted 2017-02-09; First posted 2017-02-14 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Knee Arthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- manually instrumented total knee arthroplasty (Active Comparator): Manually instrumented implantation of a total knee prosthesis involves use of cutting guides or jigs that are secured to the femur and the tibia. The femoral guide is secured to the femur after an intramedullary referenced guide is placed into the femur and the rotational alignment is then assessed with use of the epicondylar axis. An extra-medullary tibial alignment guide will be used to create the tibial cut.
  Interventions: Procedure: manually instrumented total knee arthroplasty
- robotic assisted total knee arthroplasty (Experimental): Robotically assisted surgery is used in conjunction with the preoperative CT scan and intra-operative bony registration of the patient's knee. Femoral and tibial trackers are placed and then the bone is registered using bony landmarks to allow the computer and robot to know where the patients' femur and tibia are in space. Once this is complete the preoperative templated surgical plan (performed by the PI) is used to register where to make the bony cuts in order to implant the knee components. The cutting process is performed by the surgeon with the robot assisting in guiding the cuts based on the registered CT anatomy. The surgeon has complete control of the cutting process with the assistance of the robot for placement of the cuts.
  Interventions: Device: robotic assisted total knee arthroplasty

INTERVENTIONS:
Procedure: manually instrumented total knee arthroplasty — Manually instrumented implantation of a total knee prosthesis involves use of cutting guides or jigs that are secured to the femur and the tibia. The femoral guide is secured to the femur after an intramedullary referenced guide is placed into the femur and the rotational alignment is then assessed with use of the epicondylar axis. An extra-medullary tibial alignment guide will be used to create the tibial cut.
  Arms: manually instrumented total knee arthroplasty
Device: robotic assisted total knee arthroplasty — Robotically assisted surgery is used in conjunction with the preoperative CT scan and intra-operative bony registration of the patient's knee. Femoral and tibial trackers are placed and then the bone is registered using bony landmarks to allow the computer and robot to know where the patients' femur and tibia are in space. Once this is complete the preoperative templated surgical plan (performed by the PI) is used to register where to make the bony cuts in order to implant the knee components. The cutting process is performed by the surgeon with the robot assisting in guiding the cuts based on the registered CT anatomy. The surgeon has complete control of the cutting process with the assistance of the robot for placement of the cuts.
  Arms: robotic assisted total knee arthroplasty

SUMMARY:
The purpose of this study is to compare the outcomes and accuracy of implant positioning in robotic assisted total knee arthroplasty with traditional manually instrumented total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have knee pain and are candidates for total knee arthroplasty
* Patients able to consent to be included in the study

Exclusion Criteria:

* Patients with previous total or partial knee arthroplasty in need of revision surgery
* Patients unable to or unwilling to undergo post-operative CT scans after understanding the risks and benefits

Ages: 25 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Summation of angle differences between pre-operative plan and the final implant position as indicated by computed tomography (CT) | within 2 weeks before surgery, within one month of surgery
  The absolute value of the individual differences in various angle measurements will be added together to form a total summation of angle difference.

SECONDARY OUTCOMES:
Pain as assessed by the PROMIS 10 measurement system | within 2 weeks before surgery
  Patient-Reported Outcomes Measurement Information System (PROMIS)
Pain as assessed by the PROMIS 10 measurement system | 3 months after surgery
  Patient-Reported Outcomes Measurement Information System (PROMIS)
Pain as assessed by the PROMIS 10 measurement system | 6 months after surgery
  Patient-Reported Outcomes Measurement Information System (PROMIS)
Pain as assessed by the PROMIS 10 measurement system | 1 year after surgery
  Patient-Reported Outcomes Measurement Information System (PROMIS)
Function as assessed by the PROMIS 10 measurement system | within 2 weeks before surgery
Function as assessed by the PROMIS 10 measurement system | 3 months after surgery
Function as assessed by the PROMIS 10 measurement system | 6 months after surgery
Function as assessed by the PROMIS 10 measurement system | 1 year after surgery
Knee injury and Osteoarthritis as assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS) measurement system | within 2 weeks before surgery
Knee injury and Osteoarthritis as assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS) measurement system | 3 months after surgery
Knee injury and Osteoarthritis as assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS) measurement system | 6 months after surgery
Knee injury and Osteoarthritis as assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS) measurement system | 1 year after surgery
Pain as assessed by a Visual Analogue Scale (VAS) | within 2 weeks before surgery
  Pain is rated on a scale of 0 to 10, with 10 being the highest level of pain.
Pain as assessed by a Visual Analogue Scale (VAS) | 3 months after surgery
  Pain is rated on a scale of 0 to 10, with 10 being the highest level of pain.
Pain as assessed by a Visual Analogue Scale (VAS) | 6 months after surgery
  Pain is rated on a scale of 0 to 10, with 10 being the highest level of pain.
Pain as assessed by a Visual Analogue Scale (VAS) | 1 year after surgery
  Pain is rated on a scale of 0 to 10, with 10 being the highest level of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Freedhand, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States